CLINICAL TRIAL: NCT03652740
Title: Effects of Commonly Used Medications on Mood and Choice
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB00165287; R01DA003890 (NIH)
Record Dates: First submitted 2018-08-28; First posted 2018-08-29 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Healthy
Keywords: over-the-counter; prescription medication; subjective effects
MeSH Terms: interventions — Methylphenidate; Nicotine

STUDY DESIGN:
Intervention Model Description: This is a within-subjects crossover design. This study involves administration of drug conditions in different dose sequence orders. All participants will receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Participants will be randomly assigned to one of several different dose sequences.
Who Masked: Participant, Investigator
Masking Description: Please note: This is a double-blind study. As part of instructions during the informed consent process, volunteers will be given a list of drugs they may receive rather than informing them only of the specific drugs being administered. More drugs are listed than will be administered to increase the degree to which volunteers are "blind" to the drugs being studied. Researchers will be blind to the drug conditions on any given session because a pharmacy member with no participant interaction will assign the randomized dose sequence and prepare the study drugs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Caffeine Chooser (Experimental): This is a within-subjects crossover design. Participants are not assigned to different groups/arms. All participants receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Primary outcomes will be compared between caffeine choosers and nonchoosers on Phase 3 drug conditions. Caffeine choosers and nonchoosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Interventions: Drug: Placebo; Drug: Methylphenidate; Drug: Nicotine
- Caffeine Non-Chooser (Active Comparator): This is a within-subjects crossover design. Participants are not assigned to different groups/arms. All participants receive the same drug conditions, but the order in which the participants receive the drug conditions will be different across participants. Primary outcomes will be compared between caffeine choosers and nonchoosers on Phase 3 drug conditions. Caffeine choosers and nonchoosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Interventions: Drug: Placebo; Drug: Methylphenidate; Drug: Nicotine

INTERVENTIONS:
Drug: Placebo — Capsules will contain a commonly prescribed or over-the-counter medication, or placebo. A placebo is an inactive substance that looks like the study drug, but contains no active drug.
Drug: Methylphenidate — Methylphenidate hydrochloride is administered orally at 10, 20, and 40 milligeam doses.
Drug: Nicotine — Nicotine is administered orally via capsule at 1, 2, 3 and 4 milligram doses.

SUMMARY:
This non-treatment study will examine how commonly used prescription or over-the-counter medications may influence mood and medication preference.

DETAILED DESCRIPTION:
Volunteers will participate in a double-blind study conducted over a period of about 14-17 weeks including sessions for screening, food and beverage diary review (Phase 1), drug exposure and choice sessions (Phase 2), and no-choice exposure sessions (Phase 3). During Phases 2 and 3, participants will orally ingest capsules containing varying doses of commonly prescribed over-the-counter medications and/or placebo. During screening, participants will be asked questions about participants' general characteristics including demographic information, mood, and personality. Participants will also be examined to determine medical eligibility. Eligible participants will proceed to Phase 1 in which participants will report to the laboratory to review their food and beverage intake up to three times per week and will provide saliva samples to be analyzed for caffeine content (3 sessions). During Phases 2 and 3, participants will be administered placebo or drug-containing capsules under double-blind conditions. To facilitate blindness to the study drugs being administered, caffeine, nicotine, and methylphenidate are disclosed to participants during consent among a longer list of potential drugs they may receive including other prescription and over-the-counter stimulant, sedative, and antihistamine medications. During Phase 2 (choice phase), participants will choose between caffeine (200 mg/70 kg) and placebo across 10 choice sequences. Each choice sequence consists of two exposure sessions (i.e., one session each of caffeine or placebo, order counterbalanced) and one choice session (i.e., choice between caffeine or placebo) for a total of 30 sessions in Phase 2. Following the choice phase, participants will complete the dose-effect phase (Phase 3) to measure the subjective reinforcing effects of methylphenidate (10, 20, and 40 mg/70 kg) and nicotine (1, 2, 3 and 4 mg/70 kg) under double-blind conditions. Phase 3 will consist of 13 total sessions including one session per drug/dose condition plus placebo (8 sessions), a replication of the four nicotine doses (4 sessions), and a final multiple-choice reinforcement session (1 session). During the multiple-choice reinforcement session, we will reinforce a randomly selected choice (i.e., drug vs. money) made by the participant after previous sessions as a surrogate measure of drug reinforcement. The identification of behavioral and pharmacological markers of vulnerability to the effects of drugs of abuse is important in order to inform future substance use disorder prevention and regulatory efforts.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Fluent in written and spoken English and is capable of understanding and complying with the protocol
* Medically healthy
* Non-smoker
* Appropriate dietary/over-the-counter/prescription/illicit drug use history
* Body Mass Index between 18.5 and 35
* Appropriate use of birth control in females e.g., barrier methods, hormonal contraceptives, Intra Uterine Devices (IUDs)

Exclusion Criteria:

* Known hypersensitivity to administered drugs
* Current neurological, hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary or metabolic disease for which administration of the study drugs would be contraindicated
* Current psychiatric or substance use condition that would interfere with study participation
* Diastolic blood pressure >90 mmHg or a systolic pressure of >140 mmHg
* Use of medications that would interfere with study participation
* Past prescriptions that may affect study participation
* Unwilling or unable to comply with the protocol
* Any other serious disease or condition that might affect life expectancy or make it difficult to successfully manage the subjects according to the protocol
* Females: Pregnancy, breastfeeding, or plans to become pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dustin C Lee, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Behavioral Pharmacology Research Unit, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
There is not currently a plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty five participants were enrolled in the study. Eight of the enrolled participants (4 participants phase-1, 4 participants phase-2) did not meet criteria and were not included in Phase 3. Twenty-one participants started phase 2 Choice sessions; at the conclusion of the sessions 17 participants were identified as caffeine choosers or non-choosers. Seventeen participants received the interventions in a randomized order. Participants receive each drug and each dose for only one session.
Groups:
- Dietary Monitoring: All participants (within-subject) receive the same drug conditions, but the order in which the participants receive the drug conditions will be randomized.
  Caffeine choosers, caffeine non-choosers, are identified during screening and will be randomly assigned to one of several different dose sequences.
  Caffeine choosers and non-choosers are individuals who choose caffeine or placebo during screening , respectively, 7 or more times during Phase 2 (screening).
  Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions per protocol.
- Caffeine Choice Sessions: Participants will choose between caffeine (200 mg/70 kg) and placebo.
- Caffeine Choosers: All participants (within-subject) receive the same drug conditions, but the order in which the participants receive the drug conditions will be randomized.
  Caffeine choosers, caffeine non-choosers, are identified during screening and will be randomly assigned to one of several different dose sequences.
  Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions per protocol.
- Caffeine Non-choosers: All participants (within-subject) receive the same drug conditions, but the order in which the participants receive the drug conditions will be randomized.
  Caffeine choosers and non-choosers are individuals who choose caffeine or placebo during screening , respectively, 7 or more times during Phase 2 (screening).
  Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions per protocol.
Period: Dietary Monitoring (1 Week)
Arm/Group | Dietary Monitoring | Caffeine Choice Sessions | Caffeine Choosers | Caffeine Non-choosers
Started | 25 | 0 | 0 | 0
Completed | 21 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0
Period: Caffeine Choice Sessions (Weeks 2-8)
Arm/Group | Dietary Monitoring | Caffeine Choice Sessions | Caffeine Choosers | Caffeine Non-choosers
Started | 0 | 21 | 0 | 0
Completed | 0 | 17 (21 participants started the Choice sessions. At the conclusion of the sessions, participants were identified as either caffeine choosers (8), or caffeine non-choosers (9).) | 0 | 0
Not Completed | 0 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Period: Dose Effect (Weeks 9-14)
Arm/Group | Dietary Monitoring | Caffeine Choice Sessions | Caffeine Choosers | Caffeine Non-choosers
Started | 0 | 0 | 8 | 9
Placebo | 0 | 0 | 8 | 9
10 mg Methylphenidate | 0 | 0 | 8 | 9
20 mg Methylphenidate | 0 | 0 | 8 | 9
40mg Methylphenidate | 0 | 0 | 8 | 9
1 mg Nicotine | 0 | 0 | 8 | 9
2 mg Nicotine | 0 | 0 | 8 | 9
3 mg Nicotine | 0 | 0 | 8 | 9
4 mg Nicotine | 0 | 0 | 8 | 9
Completed | 0 | 0 | 8 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study Completers
Groups:
- Caffeine Choosers; Caffeine Non-choosers: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive them is randomized.
- Total: Total of all reporting groups
Arm/Group | Caffeine Choosers | Caffeine Non-choosers | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.25 (10.02) | 28.22 (6.78) | 28.71 (8.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 3 | 4 | 7
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Participant Subjective Ratings of Drug Liking (Peak Change)
Description: Primary outcome will be peak change in participant ratings of drug liking relative to pre-drug ratings within 4 hours post-administration. Participants rate drug liking on a scale from -4 (dislike very much) to 4 (like very much) where 0 = Neutral or No Effect. This is not a treatment study, and higher or lower ratings of drug liking do not represent better or worse outcomes.
Time Frame: up to 4 hours after capsule ingestion.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Caffeine Chooser: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the interventions, but the order in which the participants receive the interventions is randomized. Outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Placebo: Capsules will contain a commonly prescribed or over-the-counter medication, or placebo. A placebo is an inactive substance that looks like the study drug, but contains no active drug.
  Methylphenidate: Methylphenidate hydrochloride is administered orally at 10, 20, and 40 milligeam doses.
  Nicotine: Nicotine is administered orally via capsule at 1, 2, 3 and 4 milligram doses.
- Caffeine Non-Chooser: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive the interventions is randomized. Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Placebo: Capsules will contain a commonly prescribed or over-the-counter medication, or placebo. A placebo is an inactive substance that looks like the study drug, but contains no active drug.
  Methylphenidate: Methylphenidate hydrochloride is administered orally at 10, 20, and 40 milligeam doses.
  Nicotine: Nicotine is administered orally via capsule at 1, 2, 3 and 4 milligram doses.
Arm/Group | Caffeine Chooser | Caffeine Non-Chooser
Number analyzed (Participants) | 8 | 9
score on a scale
  Placebo | 1.00 (1.20) | -0.11 (0.60)
  10 mg Methylphenidate | 0.88 (1.13) | 0.33 (1.31)
  20 mg Methylphenidate | 1.63 (1.19) | -0.50 (1.51)
  40 mg Methylphenidate | 1.88 (1.73) | -0.4 (1.51)
  1 mg Nicotine | 0.44 (0.94) | -0.11 (0.65)
  2 mg Nicotine | 0.44 (1.88) | -0.39 (1.02)
  3 mg Nicotine | 0.81 (1.76) | -1 (1.2)
  4 mg Nicotine | 0.5 (1.86) | -0.61 (0.78)

2. Secondary Outcome: Participant Subjective Ratings of Drug Value
Description: Secondary outcome will be subject rating of monetary drug value as assessed post-administration. Participants will rate the subjective value of the drug on a scale from -$30 (i.e., they would prefer to lose $30 rather than take the drug) to $30 (i.e., they would prefer to take today's drug instead of receiving $30). This is not a treatment study, and higher or lower ratings of drug value do not represent better or worse outcomes.
Time Frame: Completed by the participant up to 4 hours after capsule ingestion.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Caffeine Chooser; Caffeine Non-Chooser: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive the interventions is randomized. Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Placebo: Capsules will contain a commonly prescribed or over-the-counter medication, or placebo. A placebo is an inactive substance that looks like the study drug, but contains no active drug.
  Methylphenidate: Methylphenidate hydrochloride is administered orally at 10, 20, and 40 milligeam doses.
  Nicotine: Nicotine is administered orally via capsule at 1, 2, 3 and 4 milligram doses.
Arm/Group | Caffeine Chooser | Caffeine Non-Chooser
Number analyzed (Participants) | 8 | 9
units on a scale
  Placebo | 0.19 (0.81) | 0.06 (1.59)
  10 mg Methylphenidate | 0.41 (0.81) | -1.97 (12.18)
  20 mg Methylphenidate | 0.06 (3.00) | -1.14 (2.27)
  40 mg Methylphenidate | 1.34 (4.86) | 0.14 (1.91)
  1 mg Nicotine | -1.02 (2.95) | -0.42 (1.28)
  2 mg Nicotine | -2.81 (8.19) | -0.90 (2.06)
  3 mg Nicotine | -0.70 (2.35) | -4.58 (7.79)
  4 mg Nicotine | -3.09 (7.69) | -3.13 (4.02)

ADVERSE EVENTS:
Time Frame: At every study session (up to 14 weeks post enrollment)
Groups:
- Placebo: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive the interventions is randomized. Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Placebo: Capsules will contain a commonly prescribed or over-the-counter medication, or placebo. A placebo is an inactive substance that looks like the study drug, but contains no active drug.
- 10 mg Methylphenidate; 20 mg Methylphenidate; 40 mg Methylphenidate: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive the interventions is randomized. Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Methylphenidate: Methylphenidate hydrochloride is administered orally at 10, 20, and 40 milligram doses.
- 1 mg Nicotine; 2 mg Nicotine; 3 mg Nicotine; 4 mg Nicotine: This is a within-subjects crossover design. Participants are identified as caffeine choosers and caffeine non-choosers during screening. Participants in each arm will receive the same interventions, but the order in which the participants will receive the interventions is randomized. Primary outcomes will be compared between caffeine choosers and non-choosers on Phase 3 drug conditions. Caffeine choosers and non-choosers are individuals who choose caffeine or placebo, respectively, 7 or more times during Phase 2.
  Nicotine: Nicotine is administered orally via capsule at 1, 2, 3 and 4 milligram doses.
Arm/Group | Placebo | 10 mg Methylphenidate | 20 mg Methylphenidate | 40 mg Methylphenidate | 1 mg Nicotine | 2 mg Nicotine | 3 mg Nicotine | 4 mg Nicotine
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT03652740/Prot_SAP_000.pdf